CLINICAL TRIAL: NCT00578955
Title: A Randomized, Double-Masked, Parallel-Group, Comparative Study to Evaluate the Clinical and Anti-Microbial Efficacy and Safety of AzaSite Plus Compared to AzaSite Alone and Dexamethasone Alone in the Treatment of Subjects With Blepharoconjunctivitis
Brief Title: Comparative Study of AzaSite Plus Compared to AzaSite Alone and Dexamethasone Alone to Treat Subjects With Blepharoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-502-002
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Blepharoconjunctivitis
Keywords: Blepharoconjunctivitis, Ophthalmology
MeSH Terms: interventions — Azithromycin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: 1% Azithromycin and 0.1% Dexamethasone
- 2 (Active Comparator)
  Interventions: Drug: 1% Azithromycin
- 3 (Active Comparator)
  Interventions: Drug: 0.1% Dexamethasone

INTERVENTIONS:
Drug: 1% Azithromycin and 0.1% Dexamethasone — Subjects will dose topically to the eye and eyelid BID at approximately 12 hour intervals for 14 days in both eyes.
  Other Names: AzaSite Plus
  Arms: 1
Drug: 1% Azithromycin — Subjects will dose topically to the eye and eyelid BID at approximately 12 hour intervals for 14 days in both eyes.
  Other Names: AzaSite
  Arms: 2
Drug: 0.1% Dexamethasone — Subjects will dose topically to the eye and eyelid BID at approximately 12 hour intervals for 14 days in both eyes.
  Other Names: Dexamethasone
  Arms: 3

SUMMARY:
The purpose of this study is to determine if AzaSite Plus is effective and safe for the treatment of blepharoconjunctivitis compared to AzaSite alone and Dexamethasone alone.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of blepharoconjunctivitis
* Must be willing to discontinue contact lens wear for the duration of the study
* Additional inclusion criteria also apply.

Exclusion Criteria:

* Have known sensitivity or poor tolerance to any component of the study medications.
* Have any clinically significant cardiovascular disorders
* Have any history of liver or kidney disease resulting in persisting dysfunction
* Have prior (within 30 days of beginning study treatment) or anticipated concurrent use of an investigational drug or device.
* Additional exclusion criteria also apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The resolution of the clinical signs and symptoms. | 2 weeks

SECONDARY OUTCOMES:
Bacterial eradication | 2 weeks